CLINICAL TRIAL: NCT00526890
Title: Concurrent Carboplatin, Paclitaxel and Selenomethionine in Combination With Radiation for Patients With Unresectable Stage III Non-Small Cell Lung Cancer: A Phase II, Multi-Center Trial
Brief Title: Carboplatin, Paclitaxel, Selenomethionine, and Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000562780; RPCI-I-65605
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Selenomethionine; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPSR (Experimental): Concurrent Carboplatin, Paclitaxel and Selenomethionine in Combination with Radiation
  Interventions: Dietary Supplement: selenomethionine; Drug: carboplatin; Drug: paclitaxel; Other: laboratory biomarker analysis; Radiation: radiation therapy

INTERVENTIONS:
Dietary Supplement: selenomethionine — Oral Twice daily
Drug: carboplatin — Weekly IV
Drug: paclitaxel — Weekly IV
Other: laboratory biomarker analysis — Correlative Study
Radiation: radiation therapy — Undergoing radiation Therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Selenomethionine may slow the growth of tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with selenomethionine and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well selenomethionine works when given together with carboplatin, paclitaxel, and radiation therapy in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of selenomethionine in combination with chemotherapy and radiotherapy in patients with unresectable stage IIIA or IIIB non-small cell lung cancer.
* Determine if the incidence of excessive adverse events, in the form of esophagitis, pneumonitis, and myelosuppression, can be reduced with this regimen.

Secondary

* Estimate response rate, failure-free survival, and overall survival of these patients.
* Correlate selenium levels with degree of observed adverse events.

OUTLINE: This is a multicenter study.

Patients receive oral selenomethionine twice daily for 1 week and then once daily for 6 weeks. Patients also receive paclitaxel IV over 1 hour once weekly and carboplatin IV over 30 minutes once weekly for 6 weeks and undergo radiotherapy 5 days a week for 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and weekly during treatment and analyzed by absorption spectrophotometry for selenium measurement of drug concentration

After the completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), including any of the following histologic subtypes:

  * Squamous cell carcinoma
  * Adenocarcinoma (including bronchoalveolar cell carcinoma)
  * Large cell anaplastic carcinoma (including giant and clear cell carcinoma)
* Stage IIIA disease OR selected stage IIIB disease

  * T1-2, N2 disease OR T3, N2 or T4, N0-N2 disease (if based on tumor closeness to the carina, invasion of the mediastinum, or invasion of the chest wall)

    * Contralateral mediastinal disease (N3) allowed if all gross disease can be encompassed in the radiation boost field
* Tumors adjacent to a vertebral body allowed unless there is demonstrable bone invasion

  * All gross disease must be able to be encompassed in the radiation boost field
  * No direct invasion of a vertebrae body
* Unresectable or inoperable disease
* Measurable disease
* Suitable for radiotherapy, as deemed by the radiation oncologist
* No scalene, supraclavicular, or contralateral hilar node involvement
* Pleural effusion allowed provided it is transudate, cytologically negative, and non-bloody, and, according to the radiation oncologist, the tumor can be encompassed within a reasonable radiation field

  * Pleural effusion seen on chest CT scan, but not on chest x-ray, that is too small to tap is allowed
  * No exudative, bloody, or cytologically malignant effusions
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Total bilirubin ≤ 1.5 mg/dL
* Creatinine normal
* Alkaline phosphatase AND AST or ALT meeting 1 of the following criteria:

  * Alkaline phosphatase normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * Alkaline phosphatase ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * Alkaline phosphatase ≤ 5 times ULN AND AST or ALT normal
* Able to swallow oral medications
* No peripheral neuropathy > grade 1
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to selenomethionine or agents formulated with Cremophor EL
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Clinically significant cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No currently "active" second malignancy other than non-melanoma skin cancer

  * Patients are considered not to have an "active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior formal exploratory thoracotomy (N2 node identified making patient ineligible for surgery)
* No prior chemotherapy or radiotherapy for NSCLC
* No prior taxanes or platinum drugs
* No other concurrent investigational agents or anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent chemotherapy or hormonal therapy, except for the following:

  * Steroids administered for adrenal failure or septic shock
  * Hormones administered for non-disease-related conditions (e.g., insulin for diabetes)
  * Glucocorticosteroids administered as antiemetics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-10; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gomez, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPSR
Started | 16
Completed | 14
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | CPSR
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.25 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3-4 Esophagitis
Time Frame: During study treatment, up to 6 weeks
Population: Treated with Study Therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CPSR
Number analyzed (Participants) | 16
percentage of participants | 18.75 [4.05 to 45.65]

2. Primary Outcome: Incidence of Grade 3-4 Pneumonitis
Time Frame: During study treatment, up to 6 weeks
Population: Patients treated with study therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CPSR
Number analyzed (Participants) | 16
percentage of participants | 0 [0 to 20.59]

3. Primary Outcome: Incidence of Grade 3-4 Myelosuppression
Time Frame: During study treatment, up to 6 weeks
Population: Patients Treated with Study Therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CPSR
Number analyzed (Participants) | 16
percentage of participants | 12.50 [1.55 to 38.35]

4. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 month post-treatment, then q 3 months x 4
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CPSR
Number analyzed (Participants) | 16
percentage of patients | 50 [24.65 to 75.35]

5. Secondary Outcome: Failure-free Survival
Time Frame: Post-treatment follow-up every 3 months x4, then per institute standard of practice every 6 months for 2 years, then yearly therafter.
Population: Patients treated with study therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CPSR
Number analyzed (Participants) | 16
months | 9.0 [3.3 to 21.5]

6. Secondary Outcome: Overall Survival
Time Frame: as for outcome 5
Population: Patients treated with study therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CPSR
Number analyzed (Participants) | 16
months | 14.5 [7.5 to NA] — NA (not available): the upper bound of the 95% CI was not reached but is >36.4 months

7. Secondary Outcome: Selenium Level by Incidence of SAE
Description: Median Selenium level by Incidence of SAE. Mann-Whitney-Wilcoxon test was used to test the correlation between selenium levels and serious adverse events.
Time Frame: Pre-treatment and every week for 6 weeks prior to chemotherapy.
Population: All treated and eligible patients
Measure: Median (Full Range); unit: ng/mL
Arm/Group | CPSR
Number analyzed (Participants) | 16
ng/mL
  No SAE | 1435.0 [847.9 to 2870.3]
  SAE | 1803.6 [1465.0 to 2039.5]
Statistical Analysis 1: Comparison: CPSR; Mann-Whitney-Wilcoxon test was used to test the correlation between selenium levels and serious adverse events; Test type: Other; p = 0.3149, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | CPSR
Serious Adverse Events (participants affected / at risk) | 4/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPSR (N=16)
Atrial fibrillation - Grade 2 (Cardiac disorders) | 1 (1)
Oesophagitis - Grade 3 (Gastrointestinal disorders) | 1 (1)
Urinary tract infection - Grade 3 (Infections and infestations) | 1 (1)
Hypokalaemia - Grade 4 (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPSR (N=16)
Anaemia - Grade 1 (Blood and lymphatic system disorders) | 7 (9)
Anaemia - Grade 2 (Blood and lymphatic system disorders) | 4 (5)
Anaemia - Grade 3 (Blood and lymphatic system disorders) | 1 (1)
Leukopenia - Grade 1 (Blood and lymphatic system disorders) | 8 (8)
Leukopenia - Grade 2 (Blood and lymphatic system disorders) | 6 (6)
Leukopenia - Grade 3 (Blood and lymphatic system disorders) | 2 (2)
Neutropenia - Grade 1 (Blood and lymphatic system disorders) | 3 (3)
Neutropenia - Grade 2 (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia - Grade 1 (Blood and lymphatic system disorders) | 2 (2)
Arrhythmia - Grade 1 (Cardiac disorders) | 1 (1)
Tachycardia - Grade 1 (Cardiac disorders) | 2 (2)
Ear pain - Grade 2 (Ear and labyrinth disorders) | 1 (1)
Abdominal pain - Grade 1 (Gastrointestinal disorders) | 1 (1)
Abdominal pain - Grade 2 (Gastrointestinal disorders) | 1 (1)
Breath odour - Grade 1 (Gastrointestinal disorders) | 1 (1)
Chapped lips - Grade 1 (Gastrointestinal disorders) | 1 (1)
Constipation - Grade 1 (Gastrointestinal disorders) | 5 (6)
Constipation - Grade 2 (Gastrointestinal disorders) | 2 (2)
Diarrhoea - Grade 1 (Gastrointestinal disorders) | 1 (1)
Diarrhoea - Grade 2 (Gastrointestinal disorders) | 1 (1)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 2 (2)
Dyspepsia - Grade 2 (Gastrointestinal disorders) | 1 (1)
Dysphagia - Grade 1 (Gastrointestinal disorders) | 1 (1)
Nausea - Grade 1 (Gastrointestinal disorders) | 2 (2)
Nausea - Grade 2 (Gastrointestinal disorders) | 1 (1)
Oesophageal pain - Grade 2 (Gastrointestinal disorders) | 1 (1)
Oesophagitis - Grade 1 (Gastrointestinal disorders) | 5 (6)
Oesophagitis - Grade 2 (Gastrointestinal disorders) | 9 (10)
Oesophagitis - Grade 3 (Gastrointestinal disorders) | 2 (2)
Stomatitis - Grade 3 (Gastrointestinal disorders) | 1 (1)
Chest pain - Grade 1 (General disorders) | 1 (1)
Fatigue - Grade 1 (General disorders) | 6 (7)
Fatigue - Grade 2 (General disorders) | 3 (4)
Fatigue - Grade 3 (General disorders) | 1 (1)
Mucosal inflammation - Grade 2 (General disorders) | 1 (1)
Oedema peripheral - Grade 1 (General disorders) | 1 (1)
Oedema peripheral - Grade 2 (General disorders) | 1 (1)
Pain - Grade 1 (General disorders) | 1 (1)
Pain - Grade 2 (General disorders) | 2 (2)
Pyrexia - Grade 1 (General disorders) | 1 (3)
Bacterial infection - Grade 2 (Infections and infestations) | 1 (1)
Herpes zoster - Grade 2 (Infections and infestations) | 1 (1)
Infection - Grade 2 (Infections and infestations) | 1 (1)
Lower respiratory tract infection - Grade 1 (Infections and infestations) | 1 (1)
Lower respiratory tract infection - Grade 2 (Infections and infestations) | 1 (1)
Urinary tract infection - Grade 1 (Infections and infestations) | 1 (1)
Urinary tract infection - Grade 2 (Infections and infestations) | 1 (1)
Contusion - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis - Grade 2 (Injury, poisoning and procedural complications) | 3 (3)
Radiation skin injury - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Radiation skin injury - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn - Grade 1 (Injury, poisoning and procedural complications) | 2 (2)
Blood alkaline phosphatase increased - Grade 1 (Investigations) | 1 (1)
Weight decreased - Grade 1 (Investigations) | 1 (1)
Weight decreased - Grade 2 (Investigations) | 1 (1)
Anorexia - Grade 2 (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Dehydration - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia - Grade 1 (Metabolism and nutrition disorders) | 7 (10)
Hyperglycaemia - Grade 2 (Metabolism and nutrition disorders) | 5 (7)
Hyperglycaemia - Grade 3 (Metabolism and nutrition disorders) | 6 (6)
Hyperkalaemia - Grade 1 (Metabolism and nutrition disorders) | 2 (2)
Hypernatraemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia - Grade 1 (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia - Grade 1 (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia - Grade 1 (Metabolism and nutrition disorders) | 4 (4)
Arthralgia - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness - Grade 1 (Nervous system disorders) | 1 (1)
Dysgeusia - Grade 1 (Nervous system disorders) | 1 (1)
Extrapyramidal disorder - Grade 2 (Nervous system disorders) | 1 (1)
Headache - Grade 2 (Nervous system disorders) | 1 (1)
Neuropathy peripheral - Grade 1 (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy - Grade 1 (Nervous system disorders) | 1 (1)
Insomnia - Grade 2 (Psychiatric disorders) | 1 (1)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnoea - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
Deep vein thrombosis - Grade 3 (Vascular disorders) | 1 (1)
Hypotension - Grade 2 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 1 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 2 (Vascular disorders) | 1 (1)
Orthostatic hypotension - Grade 3 (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes